CLINICAL TRIAL: NCT03515018
Title: Evaluation of the Therapeutic Effect of Hydroxyurea Pulse Therapy for Chronic Myeloid Leukemia Patients
Brief Title: Evaluation of the Therapeutic Effect of HU Pulse Therapy for CML Patients
Acronym: HU
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital of Harbin Medical University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FirstAHHMU
Record Dates: First submitted 2018-04-16; First posted 2018-05-03 (Actual); Last update posted 2018-05-22 (Actual); Status verified 2017-12

CONDITIONS: Leukemia, Chronic Myeloid
Keywords: Leukemia, Myeloid, Chronic-Phase; hydroxyurea; Imatinib Mesylate; Pulse Therapy, Drug
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Leukemia, Myeloid, Chronic-Phase | interventions — Hydroxyurea; Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hydroxyurea (Experimental): Drug: hydroxyurea, pulse therapy
  Interventions: Drug: hydroxyurea
- imatinib (Active Comparator): Drug: imatinib, 400mg PO per day
  Interventions: Drug: Imatinib

INTERVENTIONS:
Drug: hydroxyurea — pulse therapy
  Other Names: HU
  Arms: Hydroxyurea
Drug: Imatinib — 400mg qd PO per day
  Other Names: Imatinib Mesylate
  Arms: imatinib

SUMMARY:
RATIONALE: Drugs used in chronic-phase chronic myelogenous leukemia (CML) aimed to avoid CML conversion (AP, BC). Hydroxyurea pulse therapy for chronic-phase CML patients is effective based on the investigator's previous studies, and the scheme cost lower than imatinib. It is not yet known the efficacy compared Hydroxyurea pulse therapy with imatinib for chronic-phase CML, especially to achieve hematological remission in short time.

PURPOSE: Non-randomized trial to compare the effectiveness of hydroxyurea pulse therapy with that of imatinib in treating chronic-phase CML patients.

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare the time of WBC decreased by 10%,20%,30%,50% of these patients treated with these two drugs. II. Compare the time of spleen size decreased by 10%,20%,30%,50% of chronic-phase chronic myelogenous leukemia patients treated with imatinib to those treated with hydroxyurea pulse therapy. III. Compare the time to achieve complete remission (CR) of these patients treated with these two drugs. iv. Estimate the overall survival, event-free survival, progression-free survival (OS, EFS, PFS) and major cytogenetic response of these patients treated with these two drugs.

OUTLINE: Patients are to receive one of two treatments. Arm I: Induction: Patients receive oral hydroxyurea daily (hydroxyurea pulse therapy) until hematological remission. Maintenance: continuing hydroxyurea pulse therapy to maintain white blood cells below 8. 0 × 109 / L. Arm II: Induction: Patients receive imatinib 400mg qd until acceptable blood counts are achieved. Maintenance: Follow the recommendations of the NCCN guidelines for chronic-phase CML treatment.

PROJECTED ACCRUAL: A total of 60 patients (30 per arm) will be accrued for this study within 2 years.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of Chronic Myelogenous Leukemia (CML) in chronic phase. Patients in either accelerated or blastic phases are not eligible.
2. No previous therapy with any drugs.
3. Age ≥ 16 years
4. Patients with uncontrolled tachyarrhythmias (such as, atrial fibrillation, paroxysmal supraventricular tachycardia, and ventricular tachycardias not adequately controlled) are not eligible.
5. Non-pregnant and non-nursing. Treatment under this protocol would expose an unborn child to significant risks. Women and men of reproductive potential should agree to use an effective means of birth control.

Exclusion Criteria:

1. Patients treated with any chemotherapy drugs.
2. Patients younger than 16 years.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-05-01 (Actual); Primary Completion 2020-05-01 (Estimated); Study Completion 2020-05-01 (Estimated)

PRIMARY OUTCOMES:
white blood cell count | 2 years
  white blood cell count decreased by 10%, 20%, 30%, 50%

SECONDARY OUTCOMES:
spleen size | 2 years
  spleen size reduced 10%, 20%, 30%, 50%
complete remission | 2 years
  the time to achieve complete remission
long-term efficacy: OS, EFS, PFS | 5 years
  OS, EFS, PFS

CONTACTS AND LOCATIONS:
Overall Officials: Jin Zhou, MD, PhD, Study Chair — First Affiliated Hospital of Harbin Medical University
Locations (1):
- the First Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang, China

REFERENCES:
- [Background] Valent P, Herndlhofer S, Schneeweiss M, Boidol B, Ringler A, Kubicek S, Gleixner KV, Hoermann G, Hadzijusufovic E, Mullauer L, Sperr WR, Superti-Furga G, Mannhalter C. TKI rotation-induced persistent deep molecular response in multi-resistant blast crisis of Ph+ CML. Oncotarget. 2017 Apr 4;8(14):23061-23072. doi: 10.18632/oncotarget.15481. PMID 28416739
- [Background] Huang J, Wang L, Chen L, Qun H, Yajing X, Fangping C, Xielan Z. Changing Treatment May Affect the Predictive Ability of European Treatment Outcome Study Scoring for the Prognosis of Patients with Chronic Myeloid Leukemia. Turk J Haematol. 2017 Mar 1;34(1):10-15. doi: 10.4274/tjh.2016.0156. Epub 2016 Oct 18. PMID 27751981